CLINICAL TRIAL: NCT04378309
Title: Illinois United: ePREP Program Evaluation
Brief Title: Illinois United ePREP Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Allen Barton, Assistant Professor, University of Illinois at Urbana-Champaign
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20837
Record Dates: First submitted 2020-05-01; First posted 2020-05-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Relationship, Marital; Relational Problems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ePrep (Experimental): The ePREP program is the online version of the Prevention and Relationship Enhancement Program. It consists of 6 self-directed online sessions and accompanying homework and brief coach calls.
  Interventions: Behavioral: ePREP

INTERVENTIONS:
Behavioral: ePREP — 6-session online psychoeducational program with supporting coach calls

SUMMARY:
The current research is designed to implement and evaluate the ePREP relationship intervention with couples throughout the state of Illinois.

DETAILED DESCRIPTION:
The objective of the research is to evaluate the effectiveness of an online intervention for help-seeking couples designed to promote individual and couple well-being. Within the United States, one-third of married couples are distressed and almost half of first marriages end in divorce/separation. Relationship distress is associated with a variety of negative health outcomes, including worsened mental and physical health problems in partners as well as internalizing and externalizing problems in children. Newly developed online intervention programs for distressed couples have shown to be efficacious, but their overall reach to the general population remains limited. The current research is designed to implement and evaluate the ePREP relationship intervention with couples throughout the state of Illinois.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Illinois
* Married, engaged, or living with their partner for at least 6 months
* Both partners willing to participate in online relationship-focused programming

Exclusion Criteria:

* One or both partners reports severe forms of intimate partner violence occurring in the relationship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2022-11-10 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction | Immediate and 6-month follow-up
  Couple Satisfaction Index
Change in Relationship Instability | Immediate and 6-month follow-up
  3 item Relationship Instability measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology)
Change in Partner Support | Immediate and 6-month follow-up
  5 item Partner Support measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology)
Change in Communication conflict | Immediate and 6-month follow-up
  4 item communication conflict measure (from Doss et al., 2020, Journal of Consulting and Clinical Psychology)
Change in Relationship confidence | Immediate and 6-month follow-up
  4 item relationship confidence measure (from Stanley et al., 1994)
Change in Intervention-target behavior | Immediate and 6-month follow-up
  PREP 3 keys (new measure created for this study, assessing participants confidence in implementing each of the 3 keys of the PREP program)

SECONDARY OUTCOMES:
Change in Partner Aggression | Immediate and 6-month follow-up
  7 item partner aggression (from Doss et al., 2020, Journal of Consulting and Clinical Psychology)
Change in Psychological distress | Immediate and 6-month follow-up
  Kessler 6 item psychological distress
Change in Anger | Immediate and 6-month follow-up
  NIH PROMIS 5 item anger measure
Change in Perceived Stress | Immediate and 6-month follow-up
  Cohen's 10 item perceived stress measure
Change in General Health | Immediate and 6-month follow-up
  SF-36 4 item general health perceptions
Change in Insomnia | Immediate and 6-month follow-up
  7 item insomnia severity index
Change in Problematic Alcohol Use | Immediate and 6-month follow-up
  PROMIS 7 item problematic alcohol use
Change in Exercise | Immediate and 6-month follow-up
  1 item exercise (CDC BRFSS 2016 adaptation)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois Extension, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No